CLINICAL TRIAL: NCT01955239
Title: Prevention of Radiation-induced Parotid Gland Dysfunction by Parotid-gland Stem-cell Sparing Intensity-modulated Radiotherapy(SCS-IMRT)
Brief Title: Parotid-gland Stem-cell Sparing Intensity-modulated Radiotherapy
Acronym: SCS-IMRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Roel Steenbakkers, M.D., Ph.D., University Medical Center Groningen
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RT2011-04
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Radiotherapy; IMRT; Stem cell; Parotid gland
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard IMRT (Active Comparator): Standard IMRT in which the mean dose to both whole parotid glands is minimized.
  Interventions: Radiation: Intensity-modulated Radiotherapy
- Stem-cell Sparing IMRT (Experimental): Stem-cell Sparing IMRT in which the mean dose to the stem cell containing region of the parotid gland is minimized
  Interventions: Radiation: Intensity-modulated Radiotherapy

INTERVENTIONS:
Radiation: Intensity-modulated Radiotherapy

SUMMARY:
Rationale:

Radiation-induced parotid gland dysfunction, often leading to xerostomia is the most-frequently occurring side-effect with a major impact on patient-reported quality of life after radiotherapy for head and neck cancer (HNC). Therefore, treatments for HNC are currently optimized to minimize the mean dose to the parotid glands. Though this resulted in a significant reduction of toxicity, 30%-40% of the patients still develop sustained parotid gland dysfunction and xerostomia.

However, in animal studies the investigators found that the dose to the sub-volume of the gland containing the parotid gland stem cells is a better predictor for dysfunction than the mean dose to the whole gland. Subsequently, this finding was confirmed in a retrospective analysis in patients. Therefore, a reduction of dose specifically in this sub-volume of the parotid glands of patients is expected to further reduce the risk of parotid gland dysfunction and xerostomia.

Objective:

To test the hypothesis that parotid gland stem cell sparing intensity modulated radiotherapy in HNC patients reduces the risk of parotid gland dysfunction and xerostomia as compared to conventional parotid gland sparing intensity modulated radiotherapy.

Study design:

Double-blind prospective randomized trial (51 patients per arm). Study population: Patients treated for tumours in the head-and-neck region with curative radiotherapy, with or without the addition of chemotherapy or cetuximab.

Intervention: Patients randomized into the experimental arm will receive a treatment in which the radiation dose to the parotid gland is re-distributed to minimize dose to the sub-volume containing the stem cells, while keeping the same mean dose to the parotid gland as a whole.

Main study parameters/endpoints:

Primary endpoint is parotid gland salivary secretion. Secondary endpoints are patient- and physician-rated xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma originating from the mucosa of the head and neck area or nasopharyngeal carcinoma originating from the nasopharynx;
* The radiotherapy includes prophylactic or therapeutic irradiation of both sides of the neck (at least level II to IV);
* Age ≥ 18 years;
* WHO performance 0-2;
* To reduce the uncertainty in the assessment of relative flow after treatment, pre-treatment parotid gland saliva production stimulated with 5% citric acid should exceed >0.1 ml/min

Exclusion Criteria:

* Postoperative radiotherapy;
* Previous radiotherapy of the head and neck region (re-irradiation);
* Unilateral radiotherapy;
* Primary salivary gland tumours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Salivary flow | 12 months after radiotherapy

SECONDARY OUTCOMES:
Patient-rated Xerostomia | 12 months after radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langendijk JA, Doornaert P, Verdonck-de Leeuw IM, Leemans CR, Aaronson NK, Slotman BJ. Impact of late treatment-related toxicity on quality of life among patients with head and neck cancer treated with radiotherapy. J Clin Oncol. 2008 Aug 1;26(22):3770-6. doi: 10.1200/JCO.2007.14.6647. PMID 18669465
- [Background] Beetz I, Schilstra C, van der Schaaf A, van den Heuvel ER, Doornaert P, van Luijk P, Vissink A, van der Laan BF, Leemans CR, Bijl HP, Christianen ME, Steenbakkers RJ, Langendijk JA. NTCP models for patient-rated xerostomia and sticky saliva after treatment with intensity modulated radiotherapy for head and neck cancer: the role of dosimetric and clinical factors. Radiother Oncol. 2012 Oct;105(1):101-6. doi: 10.1016/j.radonc.2012.03.004. Epub 2012 Apr 18. PMID 22516776
- [Background] Eisbruch A. Radiotherapy: IMRT reduces xerostomia and potentially improves QoL. Nat Rev Clin Oncol. 2009 Oct;6(10):567-8. doi: 10.1038/nrclinonc.2009.143. No abstract available. PMID 19787001
- [Background] Konings AW, Cotteleer F, Faber H, van Luijk P, Meertens H, Coppes RP. Volume effects and region-dependent radiosensitivity of the parotid gland. Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):1090-5. doi: 10.1016/j.ijrobp.2004.12.035. PMID 15990013
- [Background] Konings AW, Faber H, Cotteleer F, Vissink A, Coppes RP. Secondary radiation damage as the main cause for unexpected volume effects: a histopathologic study of the parotid gland. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):98-105. doi: 10.1016/j.ijrobp.2005.06.042. Epub 2005 Oct 13. PMID 16226398
- [Background] Lombaert IM, Brunsting JF, Wierenga PK, Faber H, Stokman MA, Kok T, Visser WH, Kampinga HH, de Haan G, Coppes RP. Rescue of salivary gland function after stem cell transplantation in irradiated glands. PLoS One. 2008 Apr 30;3(4):e2063. doi: 10.1371/journal.pone.0002063. PMID 18446241
- [Background] Lombaert IM, Brunsting JF, Wierenga PK, Kampinga HH, de Haan G, Coppes RP. Keratinocyte growth factor prevents radiation damage to salivary glands by expansion of the stem/progenitor pool. Stem Cells. 2008 Oct;26(10):2595-601. doi: 10.1634/stemcells.2007-1034. Epub 2008 Jul 31. PMID 18669914
- [Derived] Doornaert P, Dahele M, Ljumanovic R, de Bree R, Slotman BJ, Castelijns JA. Use of diffusion-weighted magnetic resonance imaging (DW-MRI) to investigate the effect of chemoradiotherapy on the salivary glands. Acta Oncol. 2015 Jul;54(7):1068-71. doi: 10.3109/0284186X.2014.987357. Epub 2014 Dec 18. No abstract available. PMID 25519706